CLINICAL TRIAL: NCT00438763
Title: Prospective Randomized Comparison: Neoprene Vs. Thermoplast Short Opponens Splinting. Outcomes After a Five-week to Sixteen-week Treatment Trial.
Brief Title: CMC Arthritis - Neoprene Vs. Thermoplast Short Opponens Splinting
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator; Director of Research, Hand Service, Massachusetts General Hospital
Other Study IDs: 2005-P-002327
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Carpometacarpal Thumb Arthritis
Keywords: CMC arthritis; splint treatment; patient satisfaction; DASH questionnaire
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Subjects using the neoprene splint.
- 2: Subjects using the orthoplast splint.

SUMMARY:
Carpometacarpal Thumb Arthritis is a disease caused by different factors and attacks mainly woman older than 50 years. The signs and symptoms consist in pain, swelling, joint instability, deformity and loss of motion. Some evidence has shown that splinting of the thumb may be of benefit. There are two methods of splinting: The first is Standard Neoprene wrap-on thumb support (in which the finger is kept in the same position with in a standard Neoprene thumb splint). The second is Thermoplast Short Opponens splint (This splint is custom-made and the thumb is use as a template to design the splint). The purpose of this study is to test and evaluate these two protocols of splinting and assess which one helps or works better in patients with thumb arthritis.

DETAILED DESCRIPTION:
Osteoarthritis of the thumb carpometacarpal joint is a common condition that affects approximately 16% to 25% of postmenopausal woman and causes pain, swelling, instability, deformity and loss of motion. This condition has been staged in 4 periods according to the degree of severity. Mild stages or stages 1 and 2 are usually treated conservatively by stabilization of the joint, which can be aggressively achieved by surgical ligament reconstruction or conservatively with thumb splints. Splinting is a typical treatment for osteoarthritis of the thumb with the goals of managing pain, stabilizing the CMC joint, and improving overall thumb function. There are limited studies showing the effectiveness of splinting for this condition indicating they are successful in decreasing pain and improving function in activities of daily living as well as radiographically improving joint stability. What is less clear is, once patients leave the clinic setting, how compliant they are with their splinting regimen. Patients with chronic illnesses tend to have compliance issues when it comes to their care. Also, there are limited studies comparing different modalities of splinting. A recent study compared custom-made short opponens thermoplastic splint with the metacarpo-phalangeal (MP) joint free to a pre-fabricated short neoprene splint. They found that patients preferred the neoprene splint but both splints provided some degree of pain relief, reduction of subluxation of the MP joint and improvement in function. Our purpose is to objectively quantify the various benefits of splinting for patients with thumb arthritis using the DASH score and assess if there is a difference between the pre-fabricated neoprene splint and the custom-made short opponens thermoplastic splint with the MP included.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older.
* Males and females diagnosed using clinical criteria as having CMC Thumb Arthritis
* Radiological diagnosis is not necessary

Exclusion Criteria:

- Patients with previous history of CMC Thumb Arthritis treated surgically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the MGH Hand and Upper Extremity service.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2005-12; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
DASH questionnaire | 6 months

SECONDARY OUTCOMES:
patient satisfaction | 6 months
pinch strength | 6 months
grip strength | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Becker SJ, Bot AG, Curley SE, Jupiter JB, Ring D. A prospective randomized comparison of neoprene vs thermoplast hand-based thumb spica splinting for trapeziometacarpal arthrosis. Osteoarthritis Cartilage. 2013 May;21(5):668-75. doi: 10.1016/j.joca.2013.02.006. Epub 2013 Feb 28. PMID 23458785